CLINICAL TRIAL: NCT03682536
Title: A Phase 3, Open-label, Randomized Study to Compare the Efficacy and Safety of Luspatercept (ACE-536) Versus Epoetin Alpha for the Treatment of Anemia Due to IPSS-R Very Low, Low or Intermediate Risk Due to Myelodysplastic Syndrome (MDS) in ESA Naïve Subjects Who Require Red Blood Cell Transfusions
Brief Title: A Study to Compare the Efficacy and Safety of Luspatercept (ACE-536) Versus Epoetin Alfa for the Treatment of Anemia Due to IPSS-R Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes (MDS) Participants Who Require Red Blood Cell Transfusions and Are ESA Naïve
Acronym: COMMANDS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-536-MDS-002; U1111-1218-1810 (Registry Identifier: WHO); 2022-501485-22 (Other: EU CTR)
Record Dates: First submitted 2018-09-07; First posted 2018-09-24 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: Luspatercept; ACE-536; Anemia; Myelodysplastic Syndromes; Blood Transfusion; RBC Transfusion; Erythropoiesis-stimulating agents; Erythropoietin; Myelodysplasia; Epoetin alpha
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia; Anemia, Refractory, with Excess of Blasts | interventions — luspatercept; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Luspatercept (Experimental)
  Interventions: Drug: Luspatercept
- Epoetin alfa (Active Comparator)
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: Luspatercept — Specified dose on specified days
  Other Names: ACE-536
  Arms: Luspatercept
Drug: Epoetin alfa — Specified dose on specified days
  Other Names: EPREX®; ERYPO®; PROCRIT®
  Arms: Epoetin alfa

SUMMARY:
The purpose of this study is to determine the effectiveness of luspatercept (ACE-536) compared to epoetin alfa on red blood cell (RBC) transfusion independence (for at least 12 weeks) with a concurrent hemoglobin increase of at least 1.5 g/dL in participants with anemia due to revised international prognostic scoring system (IPSS-R) very low, low, or intermediate risk myelodysplastic syndromes (MDS) who require RBC transfusions and have never been exposed to erythropoiesis stimulating agent (ESA).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Myelodysplastic syndromes (MDS) according to WHO 2016 classification that meets revised international prognostic scoring system (IPSS-R) classification of very low, low, or intermediate risk disease, and have < 5% blasts in bone marrow
* Endogenous serum erythropoietin (sEPO) level of < 500 U/L
* Requires Red blood cell (RBC) transfusions, as documented by the criteria: Average transfusion requirement of 2 - 6 units/8 weeks of packed red blood cells (pRBCs) confirmed for a minimum of 8 weeks immediately preceding randomization
* Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2

Exclusion Criteria:

* Clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or hypothyroidism, or any type of known clinically significant bleeding or sequestration or drug induced anemia
* Known history of diagnosis of Acute myeloid leukemia (AML)
* Uncontrolled hypertension, defined as repeated elevations of systolic blood pressure (SBP) of ≥ 150 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg despite adequate treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2027-09-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (226):
- United States (25):
  - Local Institution - 107, Berkeley, California
  - Local Institution - 115, San Diego, California
  - Local Institution - 101, Whittier, California
  - Local Institution - 104, New Haven, Connecticut
  - Local Institution - 136, Washington D.C., District of Columbia
  - Local Institution - 119, Hudson, Florida
  - Local Institution - 120, St. Petersburg, Florida
  - Local Institution - 122, Tallahassee, Florida
  - Local Institution - 108, Tampa, Florida
  - Local Institution - 118, West Palm Beach, Florida
  - Local Institution - 102, Paducah, Kentucky
  - Local Institution - 123, Bethesda, Maryland
  - Local Institution - 117, Kansas City, Missouri
  - Local Institution - 134, East Brunswick, New Jersey
  - Local Institution - 113, Hackensack, New Jersey
  - Local Institution - 105, Greenville, North Carolina
  - Local Institution - 131, Portland, Oregon
  - Univ of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Local Institution - 111, Rock Hill, South Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Local Institution - 109, Houston, Texas
  - Local Institution - 114, Salt Lake City, Utah
  - Local Institution - 132, Charlottesville, Virginia
  - Local Institution - 127, Chesapeake, Virginia
- Australia (14):
  - Local Institution - 206, Albury, New South Wales
  - Local Institution - 213, Blacktown, New South Wales
  - Local Institution - 200, Concord, New South Wales
  - Local Institution - 215, Kogarah, New South Wales
  - Local Institution - 211, Nowra, New South Wales
  - Local Institution - 210, Waratah, New South Wales
  - Local Institution - 207, Wollongong, New South Wales
  - Local Institution - 208, Auchenflower, Queensland
  - Local Institution - 202, Adelaide, South Australia
  - Local Institution - 204, Clayton, Victoria
  - Local Institution - 203, Malvern, Victoria
  - Local Institution - 209, Melbourne, Victoria
  - Local Institution - 205, West Perth, Western Australia
  - Local Institution - 212, Randwick
- Austria (2):
  - Local Institution - 442, Linz
  - Local Institution - 441, Vienna
- Belgium (7):
  - Local Institution - 475, Antwerp
  - Local Institution - 471, Brasschaat
  - Local Institution - 474, Brussels
  - Local Institution - 472, Charleroi
  - Local Institution - 473, Kortrijk
  - Local Institution - 470, Leuven
  - Local Institution - 476, Roeselare
- Canada (9):
  - Local Institution - 147, Calgary, Alberta
  - Local Institution - 145, Edmonton, Alberta
  - Local Institution - 142, Hamilton, Ontario
  - Local Institution - 140, Ottawa, Ontario
  - Local Institution - 141, Toronto, Ontario
  - Local Institution - 144, Montreal, Quebec
  - Local Institution - 148, Montreal, Quebec
  - Local Institution - 151, Saskatoon, Saskatchewan
  - Local Institution - 152, Sherbrooke
- Czechia (5):
  - Local Institution - 560, Hradec Králové
  - Local Institution - 564, Ostrava-Poruba
  - Local Institution - 563, Prague
  - Local Institution - 562, Prague
  - Local Institution - 561, Prague
- France (18):
  - Local Institution - 317, Angers
  - Local Institution - 312, Bayonne
  - Local Institution - 311, Caen
  - Local Institution - 306, La Tronche
  - Local Institution - 305, Le Mans
  - Local Institution - 309, Lille
  - Local Institution - 303, Limoges
  - Local Institution - 307, Nantes
  - Local Institution - 301, Nice
  - Local Institution - 302, Paris
  - Local Institution - 313, Paris
  - Local Institution - 308, Pessac
  - Local Institution - 315, Pierre-Bénite
  - Local Institution - 316, Poitiers
  - Local Institution - 314, Strasbourg
  - Local Institution - 300, Toulouse
  - Local Institution - 310, Tours
  - Local Institution - 304, Vandœuvre-lès-Nancy
- Germany (14):
  - Local Institution - 422, Baden-Warttemberg
  - Local Institution - 424, Berlin
  - Local Institution - 428, Cologne
  - Local Institution - 426, Dresden
  - Local Institution - 429, Duisburg
  - Local Institution - 420, Düsseldorf
  - Local Institution - 431, Hamburg
  - Local Institution - 435, Keil
  - Local Institution - 423, Koblenz
  - Local Institution - 430, Leipzig
  - Local Institution - 436, Mannheim
  - Local Institution - 421, München
  - Local Institution - 425, Winnenden
  - Local Institution - 427, Würzburg
- Greece (10):
  - Local Institution - 389, Heraklion, Irakleio
  - Local Institution - 396, Alexandroupoli
  - Local Institution - 397, Athens
  - Local Institution - 391, Athens
  - Local Institution - 395, Athens
  - Local Institution - 392, Athens
  - Local Institution - 398, Pátrai
  - Local Institution - 393, Rio Patras
  - Local Institution - 399, Thessaloniki
  - Local Institution - 390, Thessaloniki
- Hungary (3):
  - Local Institution - 535, Budapest
  - Local Institution - 534, Debrecen
  - Local Institution - 536, Nyíregyháza
- Israel (7):
  - Local Institution - 386, Haifa
  - Local Institution - 383, Jerusalem
  - Local Institution - 384, Jerusalem
  - Local Institution - 381, Kfar Saba
  - Local Institution - 385, Nahariya
  - Local Institution - 382, Tel Aviv
  - Local Institution - 380, Ẕerifin
- Italy (12):
  - Local Institution - 331, Orbassano, TO
  - Local Institution - 324, Bologna
  - Local Institution - 327, Florence
  - Local Institution - 330, Meldola
  - Local Institution - 321, Milan
  - Local Institution - 329, Padua
  - Local Institution - 326, Reggio Calabria
  - Local Institution - 328, Roma
  - Local Institution - 332, Roma
  - Local Institution - 325, Rome
  - Local Institution - 323, Rozzano
  - Local Institution - 322, Udine
- Japan (20):
  - Local Institution - 238, Matsuyama, Ehime
  - Local Institution - 244, Nagasaki, Nagasaki
  - Local Institution - 236, Sayama, Osaka
  - Local Institution - 247, Amagasaki-Shi
  - Local Institution - 249, Fujisawa-Shi
  - Local Institution - 234, Fukuoka
  - Local Institution - 237, Hitachi, Ibaraki
  - Local Institution - 231, Kamogawa
  - Local Institution - 248, Kitakyushu-Shi
  - Local Institution - 270, Nagaoka-Shi
  - Local Institution - 243, Nagoya
  - Local Institution - 235, Okayama
  - Local Institution - 242, Osaka
  - Local Institution - 241, Ōgaki
  - Local Institution - 233, Sagamihara
  - Local Institution - 246, Sapporo
  - Local Institution - 239, Sendai
  - Local Institution - 232, Shibuya-ku
  - Local Institution - 245, Shimotsuga-gun
  - Local Institution - 230, Shinagawa-ku, Tokyo
- Lithuania (2):
  - Local Institution - 540, Kaunas
  - Local Institution - 541, Vilnius
- Netherlands (5):
  - Local Institution - 462, Amsterdam
  - Local Institution - 464, Nijmegen
  - Local Institution - 460, Rotterdam
  - Local Institution - 463, Sittard-Geleen
  - Local Institution - 461, The Hague
- Poland (9):
  - Local Institution - 570, Lodz, Lódzkie
  - Local Institution - 575, Gdansk
  - Local Institution - 572, Lubin
  - Local Institution - 576, Poznan
  - Local Institution - 573, Rzwszow
  - Local Institution - 579, Słupsk
  - Local Institution - 578, Wałbrzych
  - Local Institution - 577, Wroclaw
  - Local Institution - 571, Wroclaw
- Portugal (5):
  - Local Institution - 373, Beja
  - Local Institution - 371, Braga
  - Local Institution - 372, Lisbon
  - Local Institution - 370, Porto
  - Local Institution - 374, Setúbal
- Russia (11):
  - Local Institution - 511, Kaluga
  - Local Institution - 505, Kirov
  - Local Institution - 509, Krasnoyarsk
  - Local Institution - 504, Moscow
  - Local Institution - 507, Moscow
  - Local Institution - 500, Moscow
  - Local Institution - 503, Moscow
  - Local Institution - 510, Saint Petersburg
  - Local Institution - 506, Saint Petersburg
  - Local Institution - 508, Saratov
  - Local Institution - 502, Tula
- South Korea (8):
  - Local Institution - 251, Busan
  - Local Institution - 257, Daegu
  - Local Institution - 250, Hwasun-Gun
  - Local Institution - 253, Seongnam-si
  - Local Institution - 252, Seoul
  - Local Institution - 256, Seoul
  - Local Institution - 255, Seoul
  - Local Institution - 254, Seoul
- Spain (14):
  - Local Institution - 358, Barcelona
  - Local Institution - 350, Barcelona
  - Local Institution - 354, Granada
  - Local Institution - 352, Madrid
  - Local Institution - 355, Madrid
  - Local Institution - 353, Málaga
  - Local Institution - 361, Murcia
  - Local Institution - 356, Ourense
  - Local Institution - 363, Oviedo
  - Local Institution - 362, Palma de Mallorca
  - Local Institution - 351, Salamanca
  - Local Institution - 360, Seville
  - Local Institution - 357, Valencia
  - Local Institution - 359, Valencia
- Sweden (3):
  - Local Institution - 550, Gothenburg
  - Local Institution - 552, Lund
  - Local Institution - 551, Stockholm
- Switzerland (3):
  - Local Institution - 450, Bern
  - Local Institution - 452, Lucerne
  - Local Institution - 451, Winterthur
- Taiwan (5):
  - Local Institution - 220, Changhua City, Changhua
  - Local Institution - 222, Niaosong District Kaohsiung City
  - Local Institution - 223, Taichung
  - Local Institution - 224, Taichung
  - Local Institution - 221, Taipei
- Turkey (Türkiye) (3):
  - Local Institution - 342, Ankara
  - Local Institution - 340, Manisa
  - Local Institution - 343, Trabzon
- Ukraine (6):
  - Local Institution - 526, Cherkassy
  - Local Institution - 525, Dnipro
  - Local Institution - 522, Kyiv
  - Local Institution - 520, Lviv
  - Local Institution - 523, Mykolaiv
  - Local Institution - 521, Ternopil
- United Kingdom (6):
  - Local Institution - 401, Aberdeen
  - Local Institution - 403, Bournemouth
  - Local Institution - 405, Headington, Oxford
  - Local Institution - 407, Lincoln
  - Local Institution - 404, London
  - Local Institution - 400, Manchester

REFERENCES:
- [Derived] Komrokji RS, Hayati S, Ugidos M, Garcia-Manero G, Della Porta MG, Zeidan AM, Santini V, Platzbecker U, Gandhi AK, Suragani RNVS. Impact of Mutational Landscape and Burden on RBC Transfusion Response in Patients With Lower-Risk Myelodysplastic Syndromes (LR-MDS) in the COMMANDS Study. Am J Hematol. 2026 Jan 19. doi: 10.1002/ajh.70171. Online ahead of print. PMID 41549790
- [Derived] Garcia-Manero G, Santini V, Zeidan AM, Komrokji RS, Pozharskaya V, Rose S, Keeperman K, Lai Y, Kalsekar S, Aggarwal B, Miteva D, Valcarcel D, Fenaux P, Shortt J, Della Porta MG, Platzbecker U. Long-Term Transfusion Independence with Luspatercept Versus Epoetin Alfa in Erythropoiesis-Stimulating Agent-Naive, Lower-Risk Myelodysplastic Syndromes in the COMMANDS Trial. Adv Ther. 2025 Jul;42(7):3576-3589. doi: 10.1007/s12325-025-03208-5. Epub 2025 May 16. PMID 40377899
- [Derived] Della Porta MG, Garcia-Manero G, Santini V, Zeidan AM, Komrokji RS, Shortt J, Valcarcel D, Jonasova A, Dimicoli-Salazar S, Tiong IS, Lin CC, Li J, Zhang J, Pilot R, Kreitz S, Pozharskaya V, Keeperman KL, Rose S, Prebet T, Lai Y, Degulys A, Paolini S, Cluzeau T, Fenaux P, Platzbecker U. Luspatercept versus epoetin alfa in erythropoiesis-stimulating agent-naive, transfusion-dependent, lower-risk myelodysplastic syndromes (COMMANDS): primary analysis of a phase 3, open-label, randomised, controlled trial. Lancet Haematol. 2024 Sep;11(9):e646-e658. doi: 10.1016/S2352-3026(24)00203-5. Epub 2024 Jul 19. PMID 39038479
- [Derived] Platzbecker U, Della Porta MG, Santini V, Zeidan AM, Komrokji RS, Shortt J, Valcarcel D, Jonasova A, Dimicoli-Salazar S, Tiong IS, Lin CC, Li J, Zhang J, Giuseppi AC, Kreitz S, Pozharskaya V, Keeperman KL, Rose S, Shetty JK, Hayati S, Vodala S, Prebet T, Degulys A, Paolini S, Cluzeau T, Fenaux P, Garcia-Manero G. Efficacy and safety of luspatercept versus epoetin alfa in erythropoiesis-stimulating agent-naive, transfusion-dependent, lower-risk myelodysplastic syndromes (COMMANDS): interim analysis of a phase 3, open-label, randomised controlled trial. Lancet. 2023 Jul 29;402(10399):373-385. doi: 10.1016/S0140-6736(23)00874-7. Epub 2023 Jun 10. PMID 37311468
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Luspatercept: Starting dose of 1.0 mg/kg subcutaneous injection every 3 weeks (21 days; Q3W). Dose levels can be increased in a stepwise manner beyond the starting dose to 1.33 mg/kg, and up to a maximum of 1.75 mg/kg.
- Epoetin Alfa: Starting dose of 450 IU/kg (maximum total starting dose is 40,000 IU) subcutaneous injection once every week (7 days; QW). Dose levels can be increased in a stepwise manner beyond the starting dose to 787.5 IU/kg, and up to a maximum of 1,050 IU/kg (with a maximum total dose of 80,000 IU).
Period: Randomization
Arm/Group | Luspatercept | Epoetin Alfa
Started (Randomized) | 182 | 181
Completed (Continuing to Treatment Period) | 182 | 179
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Treatment
Arm/Group | Luspatercept | Epoetin Alfa
Started | 182 | 179
Completed (Continuing in the Treatment Period) | 78 | 53
Not Completed | 104 | 126
Not completed — Other Reasons | 8 | 7
Not completed — Physician Decision | 5 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Study Terminated by Sponsor | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 16 | 18
Not completed — Lack of Efficacy | 41 | 68
Not completed — Disease Progression | 9 | 7
Not completed — Adverse Event | 9 | 5
Not completed — Death | 14 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Luspatercept | Epoetin Alfa | Total
Number analyzed (Participants) | 182 | 181 | 363
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.5 (8.92) | 73.4 (9.66) | 73.4 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 89 | 162
  Male | 109 | 92 | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 23
  Not Hispanic or Latino | 155 | 156 | 311
  Unknown or Not Reported | 16 | 13 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 25 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 146 | 143 | 289
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Red Blood Cell Transfusion Independence (RBC-TI) for 12 Weeks (84 Days) With a Mean Hemoglobin Increase ≥ 1.5 g/dL
Description: Percentage of participants who are RBC transfusion-free for any 12-week period associated with a concurrent mean hemoglobin (Hgb) increase ≥ 1.5 g/dL compared to baseline.
  After applying below 14/3-day rule, the baseline Hgb value is defined as the lowest Hgb value from the central, local laboratory, or pre transfusion Hgb from transfusion records that is within 56 days on or prior to the first dose of treatment, or randomization date if participants were not treated.
  4/3-day rule: only Hgb values that are at least 14 days after a transfusion may be used unless there is another transfusion within 3 days after the Hgb assessment. If this occurs, that Hgb value will be used despite being < 14 days after the previous transfusion.
Time Frame: Week 1 through Week 24
Population: ITT Population - all randomized participants regardless of whether or not the participant received treatment.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 181
Percent of participants | 60.4 [52.9 to 67.6] | 34.8 [27.9 to 42.2]
Statistical Analysis 1: Comparison: Luspatercept vs Epoetin Alfa; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.1, 95% CI 2-sided [2.0 to 4.8]

2. Secondary Outcome: Percentage of Participants With Red Blood Cell Transfusion Independence (RBC-TI) for 24 Weeks
Description: Red blood cell transfusion independence (RBC-TI) for 24 weeks is defined as the percentage of participants who did not receive RBC transfusions from Week 1 through Week 24.
Time Frame: Week 1 through Week 24
Population: ITT Population - all randomized participants regardless of whether or not the participant received treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 181
Percentage of participants | 47.8 [40.4 to 55.3] | 30.9 [24.3 to 38.2]
Statistical Analysis 1: Comparison: Luspatercept vs Epoetin Alfa; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.4 to 3.7]

3. Secondary Outcome: Mean Hemoglobin Change Over 24 Weeks
Description: Mean hemoglobin (Hgb) change over the 24-week period of Week 1 through Week 24 compared to baseline.
  After applying below 14/3-day rule, the baseline Hgb value is defined as the lowest Hgb value from the central, local laboratory, or pre transfusion Hgb from transfusion records that is within 56 days on or prior to the first dose of treatment, or randomization date if participants were not treated.
  4/3-day rule: only Hgb values that are at least 14 days after a transfusion may be used unless there is another transfusion within 3 days after the Hgb assessment. If this occurs, that Hgb value will be used despite being < 14 days after the previous transfusion.
Time Frame: Week 1 through Week 24
Population: ITT Population (all randomized participants regardless of whether or not the participant received treatment) with baseline measurements.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 181 | 176
g/dL | 2.0 (1.14) | 1.5 (1.12)

4. Secondary Outcome: Percentage of Participants Achieving Hematologic Improvement - Erythroid Response (HI-E) Per IWG
Description: The percentage of participants meeting the modified HI-E criteria per the International Working Group (IWG) sustained over any consecutive 56-day period in Week 1-24: For participants with baseline red blood cell (RBC) transfusion burden of >= 4 units/8 weeks, a reduction of at least 4 units RBC transfusion; for participants with baseline RBC transfusion burden of < 4 units/8 weeks, mean increase of hemoglobin of at least 1.5 g/dL in the absence of transfusions.
Time Frame: Week 1 through Week 24
Population: ITT Population - all randomized participants regardless of whether or not the participant received treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 181
Percentage of participants | 74.2 [67.2 to 80.4] | 53.0 [45.5 to 60.5]
Statistical Analysis 1: Comparison: Luspatercept vs Epoetin Alfa; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.8, 95% CI 2-sided [1.8 to 4.5]

5. Secondary Outcome: Time to Hematologic Improvement - Erythroid Response (HI-E)
Description: Time from first dose to first onset of achieving modified HI-E.
  The modified HI-E criteria per the International Working Group (IWG) sustained over any consecutive 56-day period in Week 1-24: For participants with baseline red blood cell (RBC) transfusion burden of >= 4 units/8 weeks, a reduction of at least 4 units RBC transfusion; for participants with baseline RBC transfusion burden of < 4 units/8 weeks, mean increase of hemoglobin of at least 1.5 g/dL in the absence of transfusions.
Time Frame: Week 1 through Week 24
Population: ITT Population (all randomized participants regardless of whether or not the participant received treatment) who achieve HI-E response (Week 1-24)
Measure: Median (Full Range); unit: Days
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 135 | 96
Days | 1.0 [1.0 to 113.0] | 6.0 [1.0 to 108.0]

6. Secondary Outcome: Percentage of Participants Achieving Red Blood Cell Transfusion Independence (RBC-TI) for ≥ 12 Weeks (84 Days)
Description: Percentage of participants who are RBC transfusion-free over a consecutive 84-day period.
Time Frame: Week 1 through Week 24
Population: ITT Population - all randomized participants regardless of whether or not the participant received treatment.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 181
Percent of participants | 68.1 [60.8 to 74.8] | 48.6 [41.1 to 56.1]
Statistical Analysis 1: Comparison: Luspatercept vs Epoetin Alfa; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.5, 95% CI 2-sided [1.6 to 4.0]

7. Secondary Outcome: Duration of Red Blood Cell Transfusion Independence (RBC-TI) ≥ 12 Weeks (84 Days)
Description: Maximum duration of RBC transfusion independence for participants who achieve RBC-TI ≥ 84 days.
Time Frame: Week 1 through End of Treatment (Up to approximately an average of 66 weeks and a maximum of 202 weeks)
Population: ITT Population (all randomized participants regardless of whether or not the participant received treatment) who were RBC-TI >= 12 Weeks (Week 1-24) responders
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 124 | 88
Weeks | 128.1 [108.3 to NA] — Insufficient number of participants with events | 89.7 [55.9 to 157.3]
Statistical Analysis 1: Comparison: Luspatercept vs Epoetin Alfa; Test type: Superiority; p = 0.0096, Log Rank; Hazard Ratio (HR) = 0.534, 95% CI 2-sided [0.330 to 0.864] — Calculated by Cox proportional hazard model

8. Secondary Outcome: Time to Red Blood Cell Transfusion Independence (RBC-TI) ≥ 12 Weeks (84 Days)
Description: Time from first dose to first onset of transfusion independence ≥ 84 days.
Time Frame: Week 1 through Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 124 | 88
Days | 1.0 [1.0 to 75.0] | 1.0 [1.0 to 85.0]

9. Secondary Outcome: Time to First Red Blood Cell (RBC) Transfusion
Description: Time to first RBC transfusion is defined as time from Week 1 to first RBC transfusion on treatment. Participants who maintain RBC-TI through the end of the Treatment Period or time of analysis will be censored at EOT visit date, subsequent MDS therapy start date, study discontinuation date, analysis cutoff date or death, whichever occurs first. Median is from un-stratified Kaplan-Meier method.
Time Frame: Week 1 through End of Treatment (Up to approximately an average of 66 weeks and a maximum of 202 weeks)
Population: ITT Population - all randomized participants regardless of whether or not the participant received treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 181
Days | 155.0 [80.0 to 266.0] | 42.0 [23.0 to 55.0]

10. Secondary Outcome: The Number of Red Blood Cell (RBC) Units Transfused Within the First 24 Weeks of Treatment
Description: RBC transfusion burden on treatment is defined as total number of packed red blood cell (pRBC) units transfused within the first 24 weeks of treatment since Week 1.
Time Frame: Week 1 through Week 24
Population: All participants who were randomized and received at least one dose.
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 179
RBC units | 3.8 (5.90) | 5.2 (6.36)

11. Secondary Outcome: Percentage of Participants Achieving Red Blood Cell Transfusion Independence (RBC-TI) for ≥ 56 Days (8 Weeks)
Description: Defined as percentage of participants achieving RBC-TI for >= 56 days during any consecutive 56-day period from Week 1 through Week 24.
Time Frame: Week 1 through Week 24
Population: ITT Population - all randomized participants regardless of whether or not the participant received treatment.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 181
Percent of Participants | 79.1 [72.5 to 84.8] | 64.6 [57.2 to 71.6]
Statistical Analysis 1: Comparison: Luspatercept vs Epoetin Alfa; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.4 to 3.8]

12. Secondary Outcome: Percentage of Participants Achieving Red Blood Cell Transfusion Independence (RBC-TI) for a Consecutive 24-week Period
Description: Defined as percentage of participants achieving RBC-TI for >= 168 days during any consecutive 168-day period from Week 1 through Week 48.
Time Frame: Week 1 through Week 48
Population: ITT Population (all randomized participants regardless of whether or not the participant received treatment) whose first dose date is at least 337 days from the cutoff date or discontinued early are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 163 | 167
Percent of participants | 60.7 [52.8 to 68.3] | 39.5 [32.1 to 47.4]
Statistical Analysis 1: Comparison: Luspatercept vs Epoetin Alfa; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.6, 95% CI 2-sided [1.6 to 4.3]

13. Secondary Outcome: The Number of Participants With Acute Myeloid Leukemia (AML) Progression
Description: Progression to AML is defined as a diagnosis of AML as per WHO classification of ≥ 20% blasts in peripheral blood or bone marrow.
Time Frame: From randomization to 5 years from first dose or 3 years from last dose (whichever occurs later), unless the participant withdraws consent from the study, dies or is lost to follow-up. (Up to approximately 221 weeks)
Population: ITT Population - all randomized participants regardless of whether or not the participant received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 181
Participants | 5 | 6

14. Secondary Outcome: Median Time to Acute Myeloid Leukemia (AML) Progression
Description: Time to AML progression is defined as the time between randomization and first diagnosis of AML as per WHO classification of ≥ 20% blasts in peripheral blood or bone marrow. Participants with diagnosis of AML will be considered to have had an event. Participants who have not progressed to AML at the time of analysis will be censored at the last assessment date which does not indicate progression to AML estimated by Kaplan-Meier method.
Time Frame: From randomization to first diagnosis of AML up to 5 years from first dose or 3 years from last dose (whichever occurs later), unless the participant withdraws consent from the study, dies or is lost to follow-up. (Up to approximately 221 weeks)
Population: ITT Population: all randomized participants regardless of whether or not the participant received treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 181
Months | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

15. Secondary Outcome: Overall Survival (OS)
Description: Time from date of randomization to death due to any cause
Time Frame: Randomization to death due to any cause up to 5 years from first dose or 3 years from last dose (whichever occurs later), unless the participant withdraws consent from the study, dies or is lost to follow-up. (Up to approximately 221 weeks)
Population: ITT Population - all randomized participants regardless of whether or not the participant received treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 181
Months | NA [35.3 to NA] — Insufficient number of participants with events | 42.8 [42.8 to NA] — Insufficient number of participants with events

16. Secondary Outcome: The Number of Participants With Adverse Events (AEs)
Description: Treatment-emergent adverse events include adverse events that started on or after the first dose of treatment until 42 days after the last dose of treatment, as well as those serious adverse events (SAEs) made known to the investigator at any time thereafter that are suspected of being related to treatment.
  The severity/intensity of AEs were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0). Grade 3 = Severe, Grade 4 = Life-threatening, and Grade 5 = Death.
Time Frame: From first dose to 42 days post last dose (Up to approximately an average of 72 weeks and a maximum of 208 weeks)
Population: Safety Population - all participants who were randomized and received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 182 | 179
Participants
  One TEAE | 178 | 165
  One Suspected Related TEAE | 61 | 36
  One Serious TEAE | 82 | 71
  One Suspected Related Serious TEAE | 1 | 3
  NCI CTCAE Grade 3 or 4 TEAEs | 107 | 88
  Suspected Related NCI CTCAE Grade 3 or 4 TEAEs | 14 | 4
  NCI CTCAE Grade 5 TEAE | 15 | 14
  Suspected Related NCI CTCAE Grade 5 TEAE | 1 | 0
  One TEAE Leading to Dose Interruption | 61 | 51
  One TEAE Leading to Dose Reduction | 7 | 6
  One TEAE Leading to Dose Withdrawn | 21 | 13

17. Secondary Outcome: Number of Participants With a Positive Anti-drug Antibody (ADA) Test
Description: Number of participants under each ADA positive category. A participant is counted as 'Treatment-Emergent' if there is a positive post-baseline sample while the baseline sample is ADA negative, or there is a positive post-baseline sample with a titer >= 4-fold of the baseline titer while the baseline sample is ADA positive. A participant is counted as 'Preexisting' if the baseline sample is ADA positive and the participant is not qualified for 'Treatment-Emergent'. If the participant was discontinued from study treatment earlier than one year from the first dose, additional samples will be collected if last ADA is positive.
  Baseline is defined as the last value on or before the first dose of study drug.
Time Frame: Day 1 on week 4, 10, 16, 22, and every 12 weeks (±14 days) from the 24-Week MDS Assessment visit for up to one year from the first dose
Population: Safety Population (all participants who were randomized and received at least one dose of treatment) with baseline and at least one post-baseline immunogenicity assessment result. - Luspatercept Arm Only.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept
Number analyzed (Participants) | 176
Participants
  Preexisting | 4
  Treatment-emergent | 11

18. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 is composed of 30 items that includes a global health status score ranging from: 1-7 as well as scores for 5 functional scales (physical, role, emotional, cognitive and social), 3 symptom scales (fatigue, nausea/vomiting, and pain) and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) all ranging from 1-4. Subscale scores are transformed to a 0 to 100 scale. A high score for a functional scale represents a high or healthy level of functioning; a high score for the global health status/health related quality of life (HRQoL) represents a high overall HRQoL; but a high score for a symptom scale represents a high level of symptomatology or problems. Baseline is defined as the last value on or before the first dose of study drug.
Time Frame: Baseline and week 24.
Population: All randomized participants who completed the EORTC QLQ-C30 assessment at baseline and post-baseline assessment at the respective visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 125 | 110
Score on a scale
  Global Health Status / QoL | 1.7 (16.70) | 2.7 (20.99)
  Physical Functioning | 0.1 (16.32) | 4.4 (18.30)
  Role Functioning | -1.9 (25.59) | -2.6 (26.92)
  Emotional Functioning | 2.5 (17.17) | 3.4 (18.32)
  Cognitive Functioning | 2.0 (17.79) | 0.2 (20.75)
  Social Functioning | -2.9 (20.64) | -0.9 (24.09)
  Fatigue | -1.9 (19.84) | -9.0 (23.77)
  Nausea and Vomiting | 2.1 (12.34) | -1.2 (13.11)
  Pain | -2.1 (25.40) | -1.7 (21.77)
  Dyspnea | -1.6 (22.34) | -8.8 (26.59)
  Insomnia | -4.0 (26.30) | -3.0 (33.95)
  Appetite Loss | -1.1 (23.55) | -0.0 (25.14)
  Constipation | -0.8 (21.36) | 0.9 (23.23)
  Diarrhea | 1.6 (14.58) | 1.2 (18.58)
  Financial difficulties | -0.8 (19.15) | -1.5 (22.75)

19. Secondary Outcome: Change From Baseline in the Functional Assessment of Cancer Therapy-Anemia Version 4 (FACT-An)
Description: The Functional Assessment of Cancer Therapy - Anemia (FACT-An) questionnaire includes 47 items rating on a 5-point Likert scale from 0 (not at all) to 4 (very much) (so that 0 is considered worse quality of life and 4 is good response) on five primary subscales:
  * Physical well-being (sum of 7 items, score range from 0-28)
  * Social/Family well-being (sum of 7 items, score range from 0-28)
  * Emotional well-being (sum of 6 items, score range from 0-24)
  * Functional well-being (sum of 7 items, score range from 0-28)
  * Anemia-related symptoms (sum of 20 items, score range from 0-80)
  A total score for the FACT-An can be calculated by summing the five primary subscales with a score range from 0-188. Higher scores representing better quality of life. Baseline is defined as the last value on or before the first dose of study drug.
Time Frame: Baseline, Day 1 on weeks 7,13,19, and 24.
Population: All randomized participants who completed the Fact-An assessment at baseline and post-baseline assessment at the respective visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Luspatercept | Epoetin Alfa
Number analyzed (Participants) | 145 | 133
Score on a scale
  W7D1 | 2.1 (17.41) | 3.7 (16.43)
  W13D1: number analyzed (Participants) | 136 | 121
  W13D1 | 1.8 (20.58) | 4.5 (20.36)
  W19D1: number analyzed (Participants) | 129 | 118
  W19D1 | -0.2 (19.30) | 3.1 (23.07)
  Week 24 (D169): number analyzed (Participants) | 137 | 120
  Week 24 (D169) | 1.5 (21.39) | 2.8 (22.18)

20. Secondary Outcome: Area Under the Concentration-time Curve [AUC]
Time Frame: as for outcome 17
Reporting Status: Not Posted, anticipated posting 2027-09

21. Secondary Outcome: Maximum Plasma Concentration of Drug [Cmax]
Time Frame: as for outcome 17
Reporting Status: Not Posted, anticipated posting 2027-09

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from a participants first dose to primary completion (up to approximately 221 weeks). SAEs and Other AEs were assessed from first dose to 42 days post last dose (up to approximately an average of 72 weeks and a maximum of 208 weeks).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Luspatercept | Epoetin Alfa
All-Cause Mortality (participants affected / at risk) | 39/182 | 38/181
Serious Adverse Events (participants affected / at risk) | 82/182 | 71/179
Other Adverse Events (participants affected / at risk) | 153/182 | 134/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Luspatercept (N=182) | Epoetin Alfa (N=179)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Macular hole (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 4 | 0
General physical health deterioration (General disorders) | 3 | 1
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 8 | 10
COVID-19 pneumonia (Infections and infestations) | 3 | 6
Candida pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Chronic hepatitis C (Infections and infestations) | 0 | 1
Coronavirus pneumonia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 12
Pneumonia aspiration (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 1 | 2
Suspected COVID-19 (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 4 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraganglion neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Meningorrhagia (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Prostatectomy (Surgical and medical procedures) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 1
Hypertensive urgency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Luspatercept (N=182) | Epoetin Alfa (N=179)
Anaemia (Blood and lymphatic system disorders) | 20 | 17
Neutropenia (Blood and lymphatic system disorders) | 10 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 5
Constipation (Gastrointestinal disorders) | 11 | 12
Diarrhoea (Gastrointestinal disorders) | 32 | 25
Nausea (Gastrointestinal disorders) | 25 | 15
Asthenia (General disorders) | 25 | 29
Fatigue (General disorders) | 32 | 13
Oedema peripheral (General disorders) | 26 | 14
Pyrexia (General disorders) | 9 | 11
COVID-19 (Infections and infestations) | 19 | 18
Upper respiratory tract infection (Infections and infestations) | 7 | 15
Urinary tract infection (Infections and infestations) | 14 | 7
Contusion (Injury, poisoning and procedural complications) | 4 | 10
Fall (Injury, poisoning and procedural complications) | 14 | 10
Blood creatinine increased (Investigations) | 10 | 4
Weight decreased (Investigations) | 6 | 10
Decreased appetite (Metabolism and nutrition disorders) | 10 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 9
Hyperuricaemia (Metabolism and nutrition disorders) | 12 | 10
Iron overload (Metabolism and nutrition disorders) | 2 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 16
Dizziness (Nervous system disorders) | 23 | 15
Headache (Nervous system disorders) | 20 | 15
Insomnia (Psychiatric disorders) | 11 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Hypertension (Vascular disorders) | 27 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT03682536/Prot_SAP_000.pdf